CLINICAL TRIAL: NCT01367522
Title: A Phase 1, Open-Label, Study to Evaluate Single Dose Pharmacokinetics, Safety, and Tolerability of Methylnaltrexone (MNTX) in Volunteers With Impaired Hepatic Function
Brief Title: Pharmacokinetics, Safety, and Tolerability of Methylnaltrexone in Volunteers With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, M.D., Progenics Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 1107
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Liver Dysfunction
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: SC Methylnaltrexone (MNTX)

INTERVENTIONS:
Drug: SC Methylnaltrexone (MNTX)

SUMMARY:
This is a multicenter, non-randomized, single-dose, parallel-group study. Each subject will receive a subcutaneous dose of MNTX. Eight subjects with normal hepatic function and eight subjects from each classification of hepatic impairment will be enrolled. Plasma samples will be collected before and at specified intervals after dosing and the concentration of MNTX will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18-80 years
2. Body weight greater than 100 lbs and BMI between 18-38
3. Liver values that are abnormal must not be clinically relevant as judged by the investigator. Liver enzyme and bilirubin must be less than 5 times the upper normal of reference range and may be repeated under fed conditions if abnormal. Stable hepatitis patients as well as cirrhosis patients of either etiology.

Exclusion Criteria:

1. History of current alcohol abuse with less than 1 year abstinence
2. Conditions possibly affecting drug absorption, e.g. gastrectomy or clinically significant diabetic gastroenteropathy.
3. Currently pregnant or nursing
4. Methadone use.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-03; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of SC MNTX | 20 days
  To evaluate the pharmacokinetics of MNTX administered subcutaneously as a single dose in individuals with impaired liver and hepatic function compared to healthy controls.

SECONDARY OUTCOMES:
Time of Maximum Plasma Concentration of SC MNTX | 20 days
  To evaluate the pharmacokinetics of MNTX administered subcutaneously as a single dose in individuals with impaired liver and hepatic function compared to healthy controls.
Area Under the Plasma Concentration versus Time Curve (AUC) of SC MNTX | 20 days
  To evaluate the pharmacokinetics of MNTX administered subcutaneously as a single dose in individuals with impaired liver and hepatic function compared to healthy controls.
Percentage of SC MNTX Excreted in Urine | 20 days
  To evaluate the pharmacokinetics of MNTX administered subcutaneously as a single dose in individuals with impaired liver and hepatic function compared to healthy controls.
Urinary Clearance of SC MNTX | 20 days
  To evaluate the pharmacokinetics of MNTX administered subcutaneously as a single dose in individuals with impaired liver and hepatic function compared to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States